CLINICAL TRIAL: NCT03223181
Title: Assessment of Cow's Milk-related Symptom Scoring Awareness Tool in Young Turkish Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Suna Selbuz, Assistant doctor, Ankara University
Other Study IDs: y6gyb3q8
Record Dates: First submitted 2017-05-25; First posted 2017-07-21 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Cow Milk Allergy
Keywords: Comiss
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COMİSS: Measure of CoMiSS followed by two to four weeks eviction Cow's milk protein diet and second CoMiSS measurement

SUMMARY:
In this study the investigators aimed to evaluate diagnostic accuracy the scoring tool used to determine cow's milk protein allergy, the cow's milk related symptom score, is based on the gastrointestinal, respiratory system and dermatological symptoms being together in young Turkish children.

DETAILED DESCRIPTION:
Food allergy is an immunological reaction against specific proteins in particular foods. Cow's milk protein allergy (CMPA) is a sensitivity reaction cow's milk protein via immunological pathways. CMPA is the most common food allergy under 3 years of age and its incidence is increasing in developed and developing countries. The incidence of CMPA in the first year of life is 2-3%. CMPA can be observed in breast fed, formula fed infants and infants who have started complementary food. CMPA can be classified as Ig E mediated, non Ig E mediated and mixed type according to the underlying immunological mechanisms. Basic signs and symptoms of CMPA involve the skin, gastrointestinal (GI) system and respiratory system. Ig E mediated CMPA occurs as a result of early over sensitivity to CMP and causes the clinical symptoms like urticaria, angioedema, atopic dermatitis, asthma and allergic rhinitis. Gastrointestinal symptoms like regurgitation, vomiting, colic and diarrhea may accompany. Non Ig E mediated and mixed type CMPA cause different GI signs and symptoms via inflammation and dismotility. In these groups CMPA symptoms are nonspecific like gastroesefagial reflux, regurgitation, refusal to feed , vomiting, diarrhea, bloody defecation and failure to gain weight. This type of CMPA may present as different clinical entities like protein loosing enteropathy, enterocolitis or eosinophilic eosophagitis. In some infants the only symptom can be irritability and colic.

The first step in diagnosis is a detailed clinical history and physical examination. Atopy in the patient and the family should be questioned. There is not a diagnostic test for CMPA. Serum Ig E and cow's milk specific IgE level can assist in diagnosis of CMPA in Ig E mediated CMPA however these tests are normal in non IgE mediated CMPA. The diagnosis of CMPA in suspected patients is based on the recovery of signs and symptoms with elimination of cow milk from the diet and reappearance of symptoms ad signs after challenge with cow's milk.

Nonspecific symptoms of CMPA such as regurgitation, constipation, diarrhea, and are also symptoms of functional gastrointestinal diseases in infants which are seen commonly. It has been observed that at least half of babies under 6 months experience one GI symptom. Regurgitation, colic and constipation are reported to be very common ( 23.1%, 20.5%,and 17.6%, respectively).

So the pediatricians should be aware of the fact that the symptoms or signs attributed to functional gastrointestinal diseases in infants may well be due to underlying CMPA. Therefore developing an awareness tool for pediatricians to distinguish symptoms of CMPA in infants could be useful in helping to recognize CMPA. Accurate diagnosis in affected infants ensures that infants are given appropriate diet and thus supports growth and development. On the contrary, a diet which is given without indication or continuing the diet unnecessarily after tolerance develops adversely affect growth and disturb the quality of life of the patient and the family and also cause unnecessary healthcare costs. Therefore proper recommendations and clear guidelines based on evidence are required.

In September 2014 a workshop was organized by clinicians with expertise in managing children with GI problems and atopic diseases in Brussels to review the literature and to determine benefit of a clinical score derived from symptoms associated the ingestion cow's milk proteins to primary healthcare providers. The cow's milk related symptom score (Comiss) which considers general manifestations, dermatological, gastrointestinal and respiratory system, was developed as awareness tool for cow's milk related symptoms.

This awareness tool is based on thegastrointestinal, respiratory system and dermatological symptoms being together.

This scoring tool is easy, rapid and easy to use awareness tool which pediatricians can use in determining symptoms of CMPA. It is stated that its usefulness needs to be evaluated by prospective, randomized studies.

In this prospective and randomized study the investigators aim to evaluate diagnostic accuracy using CoMISS.

Approaches and Methods to be Applied This study will include infants under 1 year of age who are admitted to Ankara University School of Medicine, Department of Pediatric Gastroenterology, Hepatology and Nutrition with GI, respiratory and dermatological symptoms and who have more than 12 points when evaluated by CoMISS. This study aims to include at least 120 patients with risk of CMPA.

Complete blood count, peripheral smear, erythrocyte sedimentation rate, albumin level, stool direct examination, occult blood in stool, Ig E and cow's milk specific IgE will be evaluated in patients who have more than 12 points according to this scoring system. At admission and follow up, symptoms and signs, physical examination findings and laboratory findings of the patients will be recorded with guidance of a form. Elimination diet to infants with a score of 12 and more will be given (elimination of cow's milk and its products from the diet of the mother in infants who are only breastfed, switching to extensively hydrolyzed formula in infants who are fed with standard formula, elimination of cow's milk and its products in infants who are fed with regular diet) for 2- 4 weeks. At the end of this period, nonresponsive infants will be switched to an amino acide based formula for 2-4 weeks .

Infants who are nonresponsive to amino acid based formula will be regarded as not having CMPA. Open cow's milk challenge test will be performed to infants who are responsive to elimination diet. After 2-4weks f elimination diet an open challenge test will e performed to infants whose findings have recovered. After this diet alteration we will confirm diagnosis of CMPA according to response of the diet. The infants in whom findings reappear after the challenge will be assessed as CMPA (+) ; while those in whom the findings don't reappear will be assessed as CMPA (-). In patients with IgE mediated CMPA, open challenge test will be performed under medical supervision in the hospital with infant formula based on cow's milk. First one drop of the infant formula will be put on infant's lips. If no reaction occurs after 15 minutes ,the infant formula based on cow's milk will be given 0.5, 1, 3, 10, 30 and 100 ml at 30-minute intervals. If no reaction occurs 2 hours after the last dosage is given, the formula will be continued at home every day with at least 200ml/day. The parents will be called by telephone to document any late reactionsIn infants with non IgE mediated CMPA , open challenge test will be performed at home Cow's milk containing foods (cake, yogurt, cheese and milk, respectively ) will be added to the mother's diet with one week intervals in exclusively breast fed infants. In formula fed infants, standart formula will be added gradually over days. In infants receiving complementary food, cooked foods containing cow's milk such as biscuit and cake will be started firstly followed by cow's milk containing foods like yogurt and cheese with 2-7 days intervals.

Predicted study duration:

- The study will be finished within 13 months.

Nature of the voluntaries:

2-weeks to 12-months-old infants admitted to outpatient clinics of Department of Pediatrics , Department of Social Pediatrics and Child Health , and Department of Gastroenterology with GI, respiratory system and/or dermatological symptoms and who have more than 12 scores in CoMİSS will be included.

ELIGIBILITY:
Inclusion Criteria:

* Reminding CMPA-respiratory system and dermatological symptoms and scoring over 12 in CoMİSS.

Exclusion Criteria:

* Infants already fed with extensive hydrolyzed formula or amino aside based on formula.
* Patients with a disease impairing normal gut transit, a known lactose intolerance severe chronic diarrhea, failure to thrive and neurological disease those that use antibiotics and those that have recently had surgical intervention or medical treatment.

Ages: 15 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients of 15 days to 1 year of age at the time of enrolment who have COMİSS score ≥12.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-06-08 (Actual); Primary Completion 2017-12-20 (Estimated); Study Completion 2017-12-25 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the cow's milk related symptom score | 8 weeks
  point change in cow's milk related symptom score within the 8 weeks follow-up period will be assess

CONTACTS AND LOCATIONS:
Overall Officials: CANSU ALTUNTAS, DR, Principal Investigator — Ankara University; ZARIFE KULOGLU, PROF, Principal Investigator — Ankara University; BETUL ULUKOL, PROF, Principal Investigator — Ankara University; SEDA TOPCU, DR, Principal Investigator — Ankara University; NISA EDA CULLAS ILARSLAN, DR, Principal Investigator — Ankara University; FATIH GUNAY, DR, Principal Investigator — Ankara University; NESLİHAN DOĞULU, MD, Principal Investigator — Ankara University
Locations (1):
- The Children's Hospital Ankara University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lifschitz C, Szajewska H. Cow's milk allergy: evidence-based diagnosis and management for the practitioner. Eur J Pediatr. 2015 Feb;174(2):141-50. doi: 10.1007/s00431-014-2422-3. Epub 2014 Sep 26. PMID 25257836
- [Background] Koletzko S, Niggemann B, Arato A, Dias JA, Heuschkel R, Husby S, Mearin ML, Papadopoulou A, Ruemmele FM, Staiano A, Schappi MG, Vandenplas Y; European Society of Pediatric Gastroenterology, Hepatology, and Nutrition. Diagnostic approach and management of cow's-milk protein allergy in infants and children: ESPGHAN GI Committee practical guidelines. J Pediatr Gastroenterol Nutr. 2012 Aug;55(2):221-9. doi: 10.1097/MPG.0b013e31825c9482. PMID 22569527
- [Background] Iacono G, Merolla R, D'Amico D, Bonci E, Cavataio F, Di Prima L, Scalici C, Indinnimeo L, Averna MR, Carroccio A; Paediatric Study Group on Gastrointestinal Symptoms in Infancy. Gastrointestinal symptoms in infancy: a population-based prospective study. Dig Liver Dis. 2005 Jun;37(6):432-8. doi: 10.1016/j.dld.2005.01.009. Epub 2005 Mar 2. PMID 15893282
- [Background] Piemontese P, Gianni ML, Braegger CP, Chirico G, Gruber C, Riedler J, Arslanoglu S, van Stuijvenberg M, Boehm G, Jelinek J, Roggero P; MIPS 1 Working Group. Tolerance and safety evaluation in a large cohort of healthy infants fed an innovative prebiotic formula: a randomized controlled trial. PLoS One. 2011;6(11):e28010. doi: 10.1371/journal.pone.0028010. Epub 2011 Nov 30. PMID 22140499
- [Result] Vandenplas Y, Dupont C, Eigenmann P, Host A, Kuitunen M, Ribes-Koninckx C, Shah N, Shamir R, Staiano A, Szajewska H, Von Berg A. A workshop report on the development of the Cow's Milk-related Symptom Score awareness tool for young children. Acta Paediatr. 2015 Apr;104(4):334-9. doi: 10.1111/apa.12902. Epub 2015 Jan 29. PMID 25557474